CLINICAL TRIAL: NCT07173179
Title: Efficacy and Safety of Papillary Epinephrine Injection Combined With Rectal Indomethacin vs Rectal Indomethacin Alone on Post ERCP Pancreatitis (PEIR-PEP): A Multi-center, Double-blind, Randomized Controlled Trial
Brief Title: Papillary Epinephrine Injection Combined With Rectal Indomethacin
Acronym: PEIR-PEP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Duzce University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Rectal NSAID vs EI combo
Record Dates: First submitted 2025-09-08; First posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Post-ERCP Acute Pancreatitis
Keywords: ERCP; post-ercp acute pancreatitis; epinephrine; indomethacin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Rectal indomethacin alone (Active Comparator): All patients in this group receive preprocedural 100mg indomethacin spp
  Interventions: Drug: Rectal indomethacin alone
- Rectal indomethacin combined wit papillary epinephrine injection (Experimental): All patients in this group receive preprocedural 100mg indomethacin spp and post-procedure 4 ml of undiluted epinephrine injected around the duodenal papilla on four quadrants, over a period of 60 seconds using a sclerotherapy needle
  Interventions: Drug: Papillary epinephrine injection combined with rectal indomethacin

INTERVENTIONS:
Drug: Papillary epinephrine injection combined with rectal indomethacin — All patients in this group receive preprocedural 100mg indomethacin spp and post-procedure 4 ml of undiluted epinephrine injected around the duodenal papilla on four quadrants, over a period of 60 seconds using a sclerotherapy needle
  Other Names: PEI
  Arms: Rectal indomethacin combined wit papillary epinephrine injection
Drug: Rectal indomethacin alone — All patients in this group receive preprocedural 100mg indomethacin spp
  Other Names: RI
  Arms: Rectal indomethacin alone

SUMMARY:
Post-endoscopic retrograde cholangiopancreatography pancreatitis (PEP) is the most common and one of the most undesirable major adverse events after endoscopic retrograde cholangiopancreatography (ERCP), causing significant morbidity and even mortality. The incidence rate is almost 15% in high-risk patients and no less than 3% in average-risk patients.

Many factors contribute to PEP, such as patient-related and endoscopist-related factors, but mainly two mechanisms are considered in terms of physiopathology: papillary edema caused by mechanical trauma during cannulation and thermal injury with electrocautery current.

Rectal NSAIDs and pancreatic stent placement are the two proven methods of PEP prophylaxis that are included in the guideline recommendations, but despite the frequent use of these methods, the incidence rates are still more than acceptable. There is a need for additional methods that are easy to implement, preferably low cost, and safe to reduce the risk of PEP.

Topical epinephrine applied submucosally can be a method that meets these goals. Ampullary epinephrine injection is an effective method in terms of post sphincterotomy bleeding but to our knowledge, there is no study examining its efficacy in PEP prophylaxis except for one retrospective study that we reported.

There are conflicting reports on epinephrine spraying on the papilla in terms of PEP, but these trials are mostly heterogeneous with different dose regimens. It should also be noted that spraying epinephrine on the papilla has a length of action of about 1 to 5 minutes but the length of action for epinephrine injection is roughly 120 minutes.

Given this information, we designed a large-scale, double-blind, randomized, controlled, superiority trial.

DETAILED DESCRIPTION:
Patient characteristics and procedure-related parameters will be recorded.

Patients will be divided into two as a patient group and a control group by 1:1 simple randomization. The patients in the indomethacin group will receive 100mg of rectal indomethacin alone, just before the procedure. In the combination group, the patients will receive 100mg of rectal indomethacin just before the procedure plus 4 quadrants of the peripapillary region will be injected with 1mL of undiluted epinephrine, 1 mL in each quadrant 1 to 2 cm away from the papillary orifice just before pulling out the duodenoscope.

The blood pressure, pulse rate, and electrocardiography will be monitored in all patients both during and after the procedure. All patients will be hospitalized for at least one night and the serum amylase and lipase levels will be measured before and again 4 hours after the procedures. Amylase, lipase, and other blood tests will also be performed routinely 24 hours after ERCP.

PEP was described as at least a threefold increase in amylase levels together with typical abdominal pain 24 hours after the procedure. Post-ERCP hyperamylasemia was defined using normal clinical conditions, but serum amylase levels were elevated above the normal upper limit (100 IU/L) 24 hours after the procedure. Patients at high risk for PEP and difficult cannulation were defined according to the European Society of Gastrointestinal Endoscopy Guidelines

ELIGIBILITY:
Inclusion Criteria:

* Patients who submitted a written informed consent for this trial, and aged between 18-80 years old
* Patients who have naïve papilla (no previous procedure was performed at ampulla)
* Patients who is suspected to have a biliary obstruction or biliary disease
* Patients who are needed to have endoscopic retrograde cholangiopancreatography for treatment of biliary obstruction

Exclusion Criteria:

* Patients who are pregnant
* Patients with mental retardation
* Patients allergic to contrast agents
* Patients who received sphincterotomy or pancreatobiliary operation previously
* Patients who have ampulla of Vater cancer
* Patients who have difficulty with the approach to ampulla due to abdominal surgery including stomach cancer with Billroth II anastomosis
* Patients who have pancreatic diseases as below (at least one more);

  * acute pancreatitis within 30days before enrollment
  * idiopathic acute recurrent pancreatitis
  * pancreas divisum
  * obstructive chronic pancreatitis
  * pancreatic cancer

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 504 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
Overall post-ERCP pancreatitis rate | 30 days
  The rate of post-ERCP pancreatitis

SECONDARY OUTCOMES:
Overall post-ERCP pancreatitis rate in high risk patients | 30 days
  The rate of post-ERCP pancreatitis in high risk patients
Overall post-ERCP hyperamylasemia | 30 days
  The rate of post-ERCP hyperamylasemia
Post sphincterotomy bleeding | 30 days
  The rate of post sphincterotomy bleeding
Overall ERCP complications | 30 days
  The rate of overall ERCP complications
Length of hospital stay | 30 days
  Days in hospital after procedure

CONTACTS AND LOCATIONS:
Overall Officials: Salih Tokmak, Principal Investigator — Duzce University
Locations (1):
- Duzce University School of Medicine, Düzce, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Andriulli A, Loperfido S, Napolitano G, Niro G, Valvano MR, Spirito F, Pilotto A, Forlano R. Incidence rates of post-ERCP complications: a systematic survey of prospective studies. Am J Gastroenterol. 2007 Aug;102(8):1781-8. doi: 10.1111/j.1572-0241.2007.01279.x. Epub 2007 May 17. PMID 17509029
- [Background] Kochar B, Akshintala VS, Afghani E, Elmunzer BJ, Kim KJ, Lennon AM, Khashab MA, Kalloo AN, Singh VK. Incidence, severity, and mortality of post-ERCP pancreatitis: a systematic review by using randomized, controlled trials. Gastrointest Endosc. 2015 Jan;81(1):143-149.e9. doi: 10.1016/j.gie.2014.06.045. Epub 2014 Aug 1. PMID 25088919
- [Background] Pezzilli R, Romboli E, Campana D, Corinaldesi R. Mechanisms involved in the onset of post-ERCP pancreatitis. JOP. 2002 Nov;3(6):162-8. PMID 12432182
- [Background] Dumonceau JM, Kapral C, Aabakken L, Papanikolaou IS, Tringali A, Vanbiervliet G, Beyna T, Dinis-Ribeiro M, Hritz I, Mariani A, Paspatis G, Radaelli F, Lakhtakia S, Veitch AM, van Hooft JE. ERCP-related adverse events: European Society of Gastrointestinal Endoscopy (ESGE) Guideline. Endoscopy. 2020 Feb;52(2):127-149. doi: 10.1055/a-1075-4080. Epub 2019 Dec 20. PMID 31863440
- [Background] Torun S, Odemis B, Cetin MF, Onmez A, Coskun O. Efficacy of Epinephrine Injection in Preventing Post-ERCP Pancreatitis. Surg Laparosc Endosc Percutan Tech. 2020 Oct 12;31(2):208-214. doi: 10.1097/SLE.0000000000000867. PMID 33048897
- [Background] Akshintala VS, Hutfless SM, Colantuoni E, Kim KJ, Khashab MA, Li T, Elmunzer BJ, Puhan MA, Sinha A, Kamal A, Lennon AM, Okolo PI, Palakurthy MK, Kalloo AN, Singh VK. Systematic review with network meta-analysis: pharmacological prophylaxis against post-ERCP pancreatitis. Aliment Pharmacol Ther. 2013 Dec;38(11-12):1325-37. doi: 10.1111/apt.12534. Epub 2013 Oct 20. PMID 24138390
- [Background] Aziz M, Ghanim M, Sheikh T, Sharma S, Ghazaleh S, Fatima R, Khan Z, Lee-Smith W, Nawras A. Rectal indomethacin with topical epinephrine versus indomethacin alone for preventing Post-ERCP pancreatitis - A systematic review and meta-analysis. Pancreatology. 2020 Apr;20(3):356-361. doi: 10.1016/j.pan.2020.02.003. Epub 2020 Feb 19. PMID 32107191
- [Background] Igawa M, Miyaoka M, Saitoh T. Influence of topical epinephrine application on microcirculatory disturbance in subjects with ulcerative colitis evaluated by laser Doppler flowmetry and transmission electron microscopy. Dig Endosc. 2000;12:126-130
- [Background] Chung SC, Leung JW, Leung FW. Effect of submucosal epinephrine injection on local gastric blood flow. A study using laser Doppler flowmetry and reflectance spectrophotometry. Dig Dis Sci. 1990 Aug;35(8):1008-11. doi: 10.1007/BF01537250. PMID 2384031